CLINICAL TRIAL: NCT05694481
Title: Effect of Circadian Rhythm Disorder on Human Intestinal Microbiota
Brief Title: An Observational Clinical Study on the Intestinal Flora in Circadian Rhythm Disorder and Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yanling Wei, Associate chief physician / Associate professor, Third Military Medical University
Other Study IDs: 20221201
Record Dates: First submitted 2022-12-13; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Circadian Rhythm Disorders; Intestinal Flora
Keywords: Circadian rhythm; Gut microbiota; Metabolomics; Metagenomes
MeSH Terms: conditions — Chronobiology Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum, feces, urine
  Serum refers to the light yellow transparent liquid separated from plasma by removing fibrinogen after blood coagulation.
  Faecalis, refers to the excretion of human and animal.
  Urine, is a fluid like metabolite excreted from the human body.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Circadian rhythm disorders: Observational, no intervention administered.
- Healthy controls: Observational, no intervention administered.

SUMMARY:
An observational clinical study on the changes of intestinal flora between people with circadian rhythm disorders and healthy controls was conducted to explore the relationship between circadian rhythm disorders and human intestinal microorganisms. To reveal the effects of circadian rhythm disorder on human intestinal microorganisms and metabolism on other potential diseases. In this study, 40 people with circadian disorders and 40 healthy controls were recruited. During the study, blood, urine and fecal samples of the subjects were obtained once, and the obtained biological samples were tested and analyzed by serum, urine metabolomics and fecal metagenomics. Subjects were also evaluated on the following scales : Circadian Type Inventory（CTI ）. The Epworth Sleeping Scale ( ESS ), Fatigue Scale-14 ( FS-14 ), Maslach Burnout Inventory-General Survey ( MBI-GS ), Athens Insomnia Scale ( AIS ), Insomnia Severity Index ( ISI ), Pittsburgh sleep quality index ( PSQI ), Bristol Stool Scale, Gastrointestinal Symptom Rating Scale ( GSRS ), Connor-Davidson resi.

DETAILED DESCRIPTION:
This study will explore the relationship between circadian rhythm disorders and human intestinal flora. The subjects were included in strict accordance with the inclusion criteria. Feces, blood, urine or other biological samples were collected and analyzed. The clinical data assessment scale and biological samples of the subjects were collected only once.

1. Data management The case report form ( CRF ) is a way of recording clinical data in clinical trials. The researchers should record all the relevant data of each subject in the experiment in a timely and true manner, and make confirmation and signature. CRF should not be changed at will. Researchers should sign and indicate the date when they do need to change. After the end of the trial, CRF was preserved by the clinical trial institution and sponsor of the researcher 's hospital. The completed CRF is reviewed by the clinical inspector and data entry is performed without modification. In order to ensure the privacy of subjects, the names of subjects on CRF need to use codes.
2. Statistical analysis The statistical analysis plan should be formulated after the finalization of the plan and finalized before the database is locked. The statistical analysis plan will specify and describe all the statistical analysis contents according to the main characteristics of the plan.
3. Preservation of data All clinical data and data analysis were recorded and managed by researchers.
4. Ethics Committee : Ethics Committee of Army Characteristic Medical Center of PLA. Application procedure : fill in the application form of ethical approval and attach the relevant approval materials.
5. Informed consent : The investigator must explain to each participant the nature, purpose, procedure, expected time, potential risks and benefits, and any discomfort that may arise, of the trial. Each subject must know that participation in the trial is voluntary and that he / she can withdraw from the trial at any time and withdraw his / her informed consent without affecting his / her subsequent treatment or relationship with the treating hysician. After explaining the basic content of the test and the researchers have been convinced that each participant will understand the purpose of the test, each participant should be required to sign the name and date on the informed consent form. Subjects should read and consider their tatements before signing and dated, and should obtain a copy of the informed consent form after signing. Subjects could not enter the trial without informed consent and without signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. All genders, Age18~75,
2. Regular night shift or day shift,
3. No antibiotics and probiotics within one month,
4. Possess understanding and communicate ability；no severe disease，no mental disorders,
5. Fully informed consent, willing to participate in this study.

Exclusion Criteria:

1. Not willing to participate in this study,
2. Patients with severe cognitive impairment or mental illness,
3. Alcohol and drug dependence,
4. The sleep disorder by alcohol and Coffee and/or Strong tea,
5. No other Tranquilizers treatment was received within 1 week before the drug was used in this clinical trial,
6. Severe intestinal infection, such as salmonella, shigella, pestis, etc,
7. Pregnant or lactating women,
8. Other reasons not suitable for clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects of the study will recruit employees with certain regularity who are engaged in night or day shifts from Daping Hospital of Army Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change of gut microbiota | Only once. The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  Alpha and Beta diversity of gut microbiota by metagenome. function and sequence-based analysis of gut microbiota microbial genome. The differential flora was obtained through differential analysis, and the correlation analysis was carried out between the differential flora and the differential metabolites. The difference in gut microbiota between people with circadian rhythm disorder and health controls is understood through stool detection.

SECONDARY OUTCOMES:
Changes in metabolites of gut microbiota | Only once.The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The comprehensive and quantitative analysis of the wide arrays of metabolites in biological samples (Fecal). After the difference metabolites are obtained through the difference analysis, the large sample data are analyzed (principal co-coordinates analysis, α/β Diversity, PLS-DA, etc.). We can more fully understand the relationship between intestinal microorganisms and circadian rhythm through metabonomic analysis.
Changes of serum metabolites | Only once.The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The comprehensive and quantitative analysis of the wide arrays of metabolites in biological samples (Serum). After the difference metabolites are obtained through the difference analysis, the large sample data are analyzed (principal co-coordinates analysis, α/β Diversity, PLS-DA, etc.). Through metabolites analysis, we can more comprehensively understand the relationship between intestinal microorganisms and circadian rhythm and blood metabolites.
Changes of urine metabolites | Only once.The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The comprehensive and quantitative analysis of the wide arrays of metabolites in biological samples (Urine). After the difference metabolites are obtained through the difference analysis, the large sample data are analyzed (principal co-coordinates analysis, α/β Diversity, PLS-DA, etc.). Through metabolites analysis, we can more comprehensively understand the relationship between intestinal microorganisms and circadian rhythm and urine metabolites.
Circadian Type Inventory | Only once.The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The amplitude and stability of their rhythms using questionnaires. (Circadian Type Inventory) CTI includes two subscales, of which the Flexibility/Rigidity scale has five items. The higher the score, the stronger the flexibility of rhythm. Languid/Vigorous has six items, and the higher the score, the more serious the fatigue of the human body.
Gastrointestinal Symptom Rating Scale (GSRS) | Only once.The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The GSRS is a brief, fairly comprehensive assessment of common gastrointestinal symptoms. The total score is 112. The higher the score, the more serious the gastrointestinal symptoms.
The Epworth Sleeping Scale（ESS） | Only once.The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The Epworth sleepiness scale (ESS) is a widely used tool which has been validated as a measure of sleepiness. The total score is 24 points. The higher the score, the more serious the sleepiness.
Fatigue Scale-14（FS-14） | Only once.The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  Evaluate the severity of people's fatigue. The total score is 14 points. The higher the score, the more fatigue.
Maslach Burnout Inventory-General Survey（MBI-GS） | Only once.The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The AIS is a self-assessment psychometric instrument designed for quantifying sleep difficulty based on the ICD-10 criteria. The total score is 21 points. The higher the score, the more serious the insomnia.
Athens Insomnia Scale（AIS） | Only once. The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The Maslach Burnout Inventory-General Survey (MBI-GS) is a widely used scale that measures burnout in the general professions. Use the standard 100 point scale for calculation. After scoring more than 50 points, the higher the score, the less positive the attitude towards work.
The Depression Anxiety Stress Scale (DASS) | Only once. The experimental group shall fill in immediately after the end of the night shift and the control group shall fill in during work. (8:00 until 12:00)
  The DASS-21 can validly be used to measure the dimensions of depression, anxiety, and stress. The total score is 63 points. The higher the score, the worse the mental state.

CONTACTS AND LOCATIONS:
Overall Officials: Yanling Wei*, MD, Principal Investigator — Daping Hospital, Army medical university
Locations (1):
- Department of Gastroenterology, Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China